CLINICAL TRIAL: NCT00217321
Title: Parkinson's Disease Registry
Brief Title: Parkinson's Disease Registry of the Muhammad Ali Parkinson Center
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Muhammad Ali Parkinson Research Center (Other)
Collaborators: Barrow Neurological Foundation (Other)
Responsible Party: Patty Hatton, CTRS/Coordinator, Barrow Neurological Institute
Other Study IDs: 03BN117
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2006-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Parkinson disease; Registry; quality of life; database
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

SUMMARY:
The purpose of the Parkinson's disease Registry is to develop a national and international database of persons with Parkinson's disease (PD). The Registry will be used to facilitate the development of new therapies and healthcare services to improve the quality of life for people with PD. It will also be a means for investigators in the field of PD to quickly identify and notify subjects about other research studies for which they are eligible.

Objectives include:

* Assess current treatment approaches and develop best-practice guidelines
* Track the functional abilities, access to healthcare and cost of illness of people with PD over time
* Drive the development of innovative research projects
* Accelerate the process of informing patients of research projects for which they may be eligible

DETAILED DESCRIPTION:
What do you need to know?

* Any individual diagnosed with PD is eligible to enroll.
* Participation in the registry is voluntary, confidential and free of charge.
* Eligible participants will be notified about opportunities to participate in clinical trials, though they are under no obligation to enter.
* Participants will need to complete an updated questionnaire every six months.
* Participants may also be asked to complete additional surveys for PD research projects.
* Any data provided will be used in scientific publications in summary form only.
* Participant names will not be released to anyone outside the Parkinson's disease Registry management team without written authorization, nor will names be sold for advertising or fund-raising purposes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease

Exclusion Criteria:

* No clinical diagnosis of Parkinson's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants must be over 18 years old, have idiopathic Parkinson's disease diagnosed by a physician.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2003-11; Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Lieberman, MD, Principal Investigator — MAPC
Locations (1):
- Muhammad Ali Parkinson Research Center, Phoenix, Arizona, United States